CLINICAL TRIAL: NCT01126866
Title: Phase II Study on Curative Resectability of Not Optimally Resectable Liver and/or Lung Metastases From Colorectal Carcinoma (CRC) Under Intensified Chemotherapy (FOLFOXIRI/ Bevacizumab)
Brief Title: Curative Resectability of Not Optimally Resectable Liver and/or Lung Metastases From Colorectal Carcinoma (CRC) Under Intensified Chemotherapy
Acronym: APRIORI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recruiting inadequate
Sponsor: National Center for Tumor Diseases, Heidelberg (Other)
Collaborators: Roche Pharma AG (Industry); Pfizer (Industry)
Responsible Party: Prof. Dr. med. Dirk Jäger, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT-2007-11-02-1003
Record Dates: First submitted 2010-05-12; First posted 2010-05-20 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-05

CONDITIONS: Colorectal Carcinoma
Keywords: advanced colorectal carcinoma; CRC; UICC Stages IV; liver and/or lung only metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- preoperative chemotherapy (Experimental)
  Interventions: Drug: intensified chemotherapy (FOLFOXIRI/Bevacizumab)

INTERVENTIONS:
Drug: intensified chemotherapy (FOLFOXIRI/Bevacizumab) — intensified chemotherapy (FOLFOXIRI/Bevacizumab)

SUMMARY:
The purpose of this clinical trial is to primarily assess the efficacy of an intensified chemotherapy consisting of a combination of FOLFOXIRI + bevacizumab. The main focus will be laid on the rate of patients who achieve secondary complete (R0)-resectable metastases.

The FOLFIRI + bevacizumab as well as the FOLFOXIRI regimens have been shown previously to be both effective in the treatment of advanced CRC with having manageable toxicities. Therefore, an intensified chemotherapy combining these two standard regimens might be a promising therapeutic approach improving the treatment of metastatic disease and outcome of CRC.

Patients with advanced colorectal carcinoma of UICC stage IV, and liver and/or lung metasta¬ses only, which are not optimally resectable, will be enrolled in this single-arm phase II study.

A minimum of 4 cycles (=8 weeks) of chemo¬therapy prior to surgery is mandatory for all patients. However, patients may withdraw from the study at any time upon their own request. Treatment with preoperative chemothera¬py will continue until 2-4 weeks prior to surgery with the last application of bevacizumab (only FOLFOXIRI) 4 weeks before surgery, at longest 16 cycles (= 32 weeks) for candidates not eli¬gible for surgery. Treatment will be discontinued prematurely at disease progression or unacceptable toxicity.

As secondary endpoints the acute and perioperative toxi¬city of preoperative chemotherapy according to NCI CTCAE v 3.0 including all peri-and post-surgical complications as well as progression free survival and overall survival and quality of life will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Indication:

   * Histologically confirmed advanced colorectal carcinoma of UICC Stages IV with liver and/or lung only metastases,which are not optimally resectable
   * Measurable disease according to RECIST criteria.
   * In case of liver metastases: 70% liver replacement and/or > 6 segments tumor involved, and/or involvement of all three hepatic veins, and/or involvement of the right and left portal pedicle, and/ or involvement of the vena cava.
   * In case of lung metastases: No tumor with direct infiltration of myocardium, esophagus, spine or intrapericardial large vessels. Preoperative data indicate a significant loss of pulmonary function after pulmonary metastasectomy with severe impairment of quality of life.
3. ECOG performance status of < 2.
4. Life expectancy of > 3 months
5. Laboratory parameters:

   * Proteinuria at baseline:

     * Patients with proteinuria <2+ on dipstick urinalysis.
     * Patients with 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-h urine collection and must have proteinuria <= 1 g of protein/24 h.
   * The required laboratory values at baseline are as follows:

     * Hematology:

       * Absolute neutrophil count (ANC) > 1.5 x 109/L
       * Platelet count > 100 x 109/L
       * Hemoglobin > 9 g/dL (may be transfused to maintain or exceed this level)
       * International Normalized Ratio (INR) < 1.5; aPTT <1.5 x ULN
     * Biochemistry:

       * Total bilirubin < 1.5 x upper limit of normal (ULN)
       * AST, ALT < 2.5 x ULN in patients without liver metastases; < 5 x ULN in patients with liver metastases
       * Serum creatinine <2.0 mg/dL or 177 ƒÝmol/L
6. Willingness to give written informed consent, written consent for data protection and willingness to participate and to comply with the study.

Exclusion Criteria:

1. Past or current history of malignancies other than colorectal carcinoma. Patients with curatively treated basal and squamous cell carcinoma of the skin and/or in-situ carcinoma of the cervix are eligible.
2. Previous chemotherapy (except adjuvant chemotherapy).
3. Extrahepatic and/or extrapulmonary meta-stases except of the initially removed lymph node metastases.
4. History or evidence upon physical examination of CNS disease unless adequately treated (e.g., seizure not controlled with standard medical therapy or history of stroke).
5. Major surgical procedures, open biopsy, or significant traumatic injury within 28 days prior to study treatment start (wound healing has to be completed), or anticipation of the need for major surgical procedure during the course of the study.
6. Evidence of bleeding diathesis or coagulopathy
7. Serious, non-healing wound, ulcer, or bone fracture
8. Treatment with investigational agents or participation in clinical trials within 30 days before study entry.
9. Clinically significant (i.e. active) cardiovascular disease, e.g., uncontrolled hyper-tension, cerebrovascular accidents (. 6 months prior to treatment start), myocardial infarction (. 6 months prior to treatment start), unstable angina, New York Heart Association (NYHA) grade . II, congestive heart failure, serious cardiac arrhythmia requiring medication.
10. Current or recent serious polyneuropathy (grade . 1 according to NCI CTCAE v3.0 criteria; exception: absence of tendon reflexes)
11. Hematopoietic diseases.
12. Known intra-abdominal inflammatory pro-cess or serious gastrointestinal ulceration.
13. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
14. Thromboembolic events or severe hemorrhage ("T 6 months before treatment start).
15. Known hypersensitivity to oxaliplatin, the background medication (bevacizumab, FA or 5-FU) or to their compounds, incl. Chinese hamster ovary (CHO) cell proteins or other recombinant human or humanized antibodies.
16. Known Gilbert-Syndrome
17. Evidence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational regimen or patient at high risk from treatment complications
18. As the following medication(s) can have interactive effects and may interfere with the patient's ability to meet the study requirements, they cannot be administered during the clinical study:

    * sorivudine or analog compounds.
    * Current or recent (within 10 days of first dose of study treatment) treatment with full-dose oral or parenteral anticoagulants or thrombolytic agents (e.g., marcumar therapy) for therapeutic purposes.
    * Current or recent (within 10 days of first dose of study treatment) chronic use of aspirin (> 325 mg/day) or clopidogrel (> 75 mg/day).
19. Women, lactating, pregnant or of child-bearing potential and fertile men not using a highly effective contraceptive method1.

    [Women of childbearing potential must have a negative pregnancy test (serum b-HCG) within 7 days before the first dose of study drug].
20. Patients who are confined by order of either judicial or administrative authorities (according to ¡± 40 Abs. 1 S. 3 AMG).
21. Patients who are incapable to understand the aim, importance and consequences of the study and to give legal informed consent (according to ¡± 40 Abs. 4 and ¡± 41 Abs. 2 and Abs. 3 AMG).
22. Patients with a history of a psychological illness or condition such as to interfere with the patient's ability to understand the requirements of the study.
23. Patients who possibly are dependent on the sponsor or investigator.
24. Patients who have participated in this study before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
surgically complete resectability; S-CR | 12 month after Surgery
  To evaluate the proportion of patients who achieve surgically complete resectability (S-CR) of metastases after preoperative chemotherapy.

SECONDARY OUTCOMES:
Evaluate the acute and perioperative toxicity of preoperative chemotherapy according to NCI CTCAE v3.0 and all peri-and post-surgical complications | 12 month after surgery
  Descriptive analysis is performed to identify treatment side effects and their individual impact from the patients' perspective, as well as changes during treatment based on BELISPO questionnaire data.
Survival rate (OS) and progression free survival (PFS) | 12 months after surgery or end of treatment.
  The PFS is calculated for all patients. It is defined as the time from admission to the study to objective tumor progression or death from any cause, whichever occurs first. OS is defined as the time from registration to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Jaeger, Prof. Dr., Study Director — NCT Heidelberg
Locations (1):
- NCT, Heidelberg, Germany